CLINICAL TRIAL: NCT02824692
Title: The Incidence of Significant Clinical Findings Using Focused Ultrasound Examination for the Heart, Lungs and Abdomen in Elderly Patients Before Emergent Surgery
Brief Title: Preoperative Significant Clinical Findings Using Focused Ultrasound Examination
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dekel Lait MD, Dr., Rambam Health Care Campus
Other Study IDs: 0117-16-RMBCTIL
Record Dates: First submitted 2016-06-18; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: heart lungs and abdomen ultrasound
  Other Names: VIVID5S GE device

SUMMARY:
The purpose of this study is to determine whether a focused ultrasound examination for the heart, lungs and abdomen, preformed by a trained anesthesiologist, can reveal significant clinical findings in elderly patients before emergent surgery.

DETAILED DESCRIPTION:
Emergent orthopedic and urological surgeries in the elderly population are characterized by high incidence of chronic diseases of the target population on one hand, and the time factor which limits the possibility to properly assess the preoperative condition on the other hand.

Therefore, anesthesiologist often perform these procedures such as hip replacement with insufficient data as compared to an elective case.

In Israel, a hip fracture must be operated on within 18 hours. This type of fracture is common to the elderly population who naturally suffer more from chronic diseases that might influence the management of anesthesia. Due to the emergent nature of the procedures involved, the patients are often operated on with only basic preoperative assessment such as ECG, chest x-ray and blood tests.

A more elaborated assessment, such as a valid echocardiography , evaluation of pleural effusion or the presence of ascites are often impossible to acquire due to inaccessibility of the echo lab (high burden, missing qualified personal ) or the availability of operation theater.

This is an observational pilot study in which the ability of a focused, bedside preoperative ultrasound examination preformed by a qualified anesthesiologist to expose significant clinical data will be evaluated.

Sample size: 30 patient. Male and female over the age 65. The examination will cover the heart (eg. volemic status, global systolic function, existence of severe valvular pathology, pericardial effusion), lungs (eg. pleural effusion, atelectasis, pneumothorax ) and abdomen ( e.g ascites ). It will be preformed at the patient bed using the VIVID5S General Electric device. All fields will be examined using the low frequency cardiac probe.

The data will be documented and saved electronically by the main investigator. All recorded ultrasound examination will be saved and coded with a number (no patient details).

All data collected will be validated by a physician experienced in the field. Any mismatch between the anesthesiologist records to the validated data will be documented.

Clinically significant findings will be documented and transferred (after validation) to the anesthesiologist performing the anesthesia (only senior anesthesiologist ).

On the following day, the anesthesiologist will document :

1. Any changes in anesthetic management due to the examination findings
2. Subjective report regarding the utility of the examination

Anesthetic changes and subjective report will be graphically documented. The anesthesiologist preforming the examination underwent the necessary qualifications to preform the exam. In any case, the preoperative examination and operation will not be held by the same anesthesiologist.

Patient enrollment to the study will be preformed at the ward, E.R or preoperative hall. It must be emphasized that in any case the performance of the operation will not be detained by the examination.

ELIGIBILITY:
Inclusion Criteria:

* male and female over 65 years
* emergent operation (within 72 hours)
* No echocardiographic examination in the past 6 months

Exclusion Criteria:

* echocardiographic examination in the past 6 months
* examination will detain surgery
* unstable patients
* no legal guardian, not eligible for informed consent
* poor ultrasound image

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly male and female (over 65 years old) undergoing emergent (within 24 -72 hours from diagnosis) orthopedic or urological procedure.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of significant clinical findings using focused ultrasound examination for the heart, lungs and abdomen in elderly patients before emergent surgery | up to 55 weeks
  Clinical findings that are considered significant (eg. pneumothorax, severe aortic stenosis, pericardial effusion) will be documented and presented in a table - demonstrating their prevalence among the study population.

SECONDARY OUTCOMES:
Sensitivity and specificity of a qualified anesthesiologist in the diagnosis of clinically significant findings in focused ultra sound examination for the heart, lung and abdoman | up to 55 weeks
  Significant clinical finding that will be missed or wrongly diagnosed by the anesthesiologist will be noted
Changes in anesthetic management following the focused ultrasound examination | up to 55 weeks
  The data will be collected and presented in a table stressing the changes made and their prevalence in the study population
Overall satisfaction of anesthesiologists from the clinical data provided to them | up to 55 weeks
  The data will be collected through a questionnaire containing numerical answers (between 1-5) regarding the usefulness and credibility of the ultra sound exam

CONTACTS AND LOCATIONS:
Overall Officials: lior fuchs, MD, Study Director — Soroka University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barber RL, Fletcher SN. A review of echocardiography in anaesthetic and peri-operative practice. Part 1: impact and utility. Anaesthesia. 2014 Jul;69(7):764-76. doi: 10.1111/anae.12663. Epub 2014 Apr 28. PMID 24773366
- [Background] Canty DJ, Royse CF, Kilpatrick D, Williams DL, Royse AG. The impact of pre-operative focused transthoracic echocardiography in emergency non-cardiac surgery patients with known or risk of cardiac disease. Anaesthesia. 2012 Jul;67(7):714-20. doi: 10.1111/j.1365-2044.2012.07118.x. Epub 2012 Mar 27. PMID 22452367
- [Background] Kertai MD, Bountioukos M, Boersma E, Bax JJ, Thomson IR, Sozzi F, Klein J, Roelandt JR, Poldermans D. Aortic stenosis: an underestimated risk factor for perioperative complications in patients undergoing noncardiac surgery. Am J Med. 2004 Jan 1;116(1):8-13. doi: 10.1016/j.amjmed.2003.07.012. PMID 14706659
- [Background] Subramani S, Tewari A. Pre-operative echocardiography: Evidence or experience based utilization in non-cardiac surgery? J Anaesthesiol Clin Pharmacol. 2014 Jul;30(3):313-5. doi: 10.4103/0970-9185.137258. No abstract available. PMID 25190935
- [Background] Oren-Grinberg A, Talmor D, Brown SM. Focused critical care echocardiography. Crit Care Med. 2013 Nov;41(11):2618-26. doi: 10.1097/CCM.0b013e31829e4dc5. PMID 23989172
- [Background] Jasudavisius A, Arellano R, Martin J, McConnell B, Bainbridge D. A systematic review of transthoracic and transesophageal echocardiography in non-cardiac surgery: implications for point-of-care ultrasound education in the operating room. Can J Anaesth. 2016 Apr;63(4):480-7. doi: 10.1007/s12630-015-0524-7. Epub 2015 Oct 30. PMID 26514983
- [Background] Michelena HI, Abel MD, Suri RM, Freeman WK, Click RL, Sundt TM, Schaff HV, Enriquez-Sarano M. Intraoperative echocardiography in valvular heart disease: an evidence-based appraisal. Mayo Clin Proc. 2010 Jul;85(7):646-55. doi: 10.4065/mcp.2009.0629. PMID 20592170
- [Background] Canty DJ, Royse CF, Kilpatrick D, Bowyer A, Royse AG. The impact on cardiac diagnosis and mortality of focused transthoracic echocardiography in hip fracture surgery patients with increased risk of cardiac disease: a retrospective cohort study. Anaesthesia. 2012 Nov;67(11):1202-9. doi: 10.1111/j.1365-2044.2012.07300.x. Epub 2012 Sep 5. PMID 22950446
- [Background] Canty DJ, Royse CF. Audit of anaesthetist-performed echocardiography on perioperative management decisions for non-cardiac surgery. Br J Anaesth. 2009 Sep;103(3):352-8. doi: 10.1093/bja/aep165. Epub 2009 Jun 23. PMID 19549642
- [Background] Luttrell K, Nana A. Effect of Preoperative Transthoracic Echocardiogram on Mortality and Surgical Timing in Elderly Adults with Hip Fracture. J Am Geriatr Soc. 2015 Dec;63(12):2505-2509. doi: 10.1111/jgs.13840. Epub 2015 Dec 11. PMID 26659463
- [Background] Canty DJ, Royse CF, Kilpatrick D, Bowman L, Royse AG. The impact of focused transthoracic echocardiography in the pre-operative clinic. Anaesthesia. 2012 Jun;67(6):618-25. doi: 10.1111/j.1365-2044.2012.07074.x. Epub 2012 Feb 21. PMID 22352785
- [Background] Alsaddique A, Royse AG, Royse CF, Mobeirek A, El Shaer F, AlBackr H, Fouda M, Canty DJ. Repeated Monitoring With Transthoracic Echocardiography and Lung Ultrasound After Cardiac Surgery: Feasibility and Impact on Diagnosis. J Cardiothorac Vasc Anesth. 2016 Apr;30(2):406-12. doi: 10.1053/j.jvca.2015.08.033. Epub 2015 Aug 29. PMID 26723882
- [Background] Ng A, Swanevelder J. Perioperative echocardiography for non-cardiac surgery: what is its role in routine haemodynamic monitoring? Br J Anaesth. 2009 Jun;102(6):731-4. doi: 10.1093/bja/aep100. No abstract available. PMID 19451153
- [Background] Loxdale SJ, Sneyd JR, Donovan A, Werrett G, Viira DJ. The role of routine pre-operative bedside echocardiography in detecting aortic stenosis in patients with a hip fracture. Anaesthesia. 2012 Jan;67(1):51-54. doi: 10.1111/j.1365-2044.2011.06942.x. Epub 2011 Oct 24. PMID 22023667
- [Background] 15. Israel Ministry of health, guidelines for quality measurements 2016, pages 25-27
- [Background] Bernier-Jean A, Albert M, Shiloh AL, Eisen LA, Williamson D, Beaulieu Y. The Diagnostic and Therapeutic Impact of Point-of-Care Ultrasonography in the Intensive Care Unit. J Intensive Care Med. 2017 Mar;32(3):197-203. doi: 10.1177/0885066615606682. Epub 2016 Jul 9. PMID 26423745
- [Background] Mantuani D, Frazee BW, Fahimi J, Nagdev A. Point-of-Care Multi-Organ Ultrasound Improves Diagnostic Accuracy in Adults Presenting to the Emergency Department with Acute Dyspnea. West J Emerg Med. 2016 Jan;17(1):46-53. doi: 10.5811/westjem.2015.11.28525. Epub 2016 Jan 12. PMID 26823930
- [Background] Piette E, Daoust R, Denault A. Basic concepts in the use of thoracic and lung ultrasound. Curr Opin Anaesthesiol. 2013 Feb;26(1):20-30. doi: 10.1097/ACO.0b013e32835afd40. PMID 23103845
- [Background] Lee CW, Kory PD, Arntfield RT. Development of a fluid resuscitation protocol using inferior vena cava and lung ultrasound. J Crit Care. 2016 Feb;31(1):96-100. doi: 10.1016/j.jcrc.2015.09.016. Epub 2015 Sep 25. PMID 26475100
- [Background] Zieleskiewicz L, Muller L, Lakhal K, Meresse Z, Arbelot C, Bertrand PM, Bouhemad B, Cholley B, Demory D, Duperret S, Duranteau J, Guervilly C, Hammad E, Ichai C, Jaber S, Langeron O, Lefrant JY, Mahjoub Y, Maury E, Meaudre E, Michel F, Muller M, Nafati C, Perbet S, Quintard H, Riu B, Vigne C, Chaumoitre K, Antonini F, Allaouchiche B, Martin C, Constantin JM, De Backer D, Leone M; CAR'Echo and AzuRea Collaborative Networks. Point-of-care ultrasound in intensive care units: assessment of 1073 procedures in a multicentric, prospective, observational study. Intensive Care Med. 2015 Sep;41(9):1638-47. doi: 10.1007/s00134-015-3952-5. Epub 2015 Jul 10. PMID 26160727